CLINICAL TRIAL: NCT01280318
Title: Profile of Plasma Growth Factors Before and After Head and Neck Oncological or Non-oncological Surgery
Acronym: HNSCC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL-ONCO 2008-03; Academic study
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Growth Factor; Surgery
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): patients with operable head and neck squamous cell carcinoma
  Interventions: Procedure: head and neck surgery
- 2 (Other): patients treated by neck ansd head surgery for a non-oncological disease
  Interventions: Procedure: head and neck surgery
- 3 (Experimental): patients treated before surgery with 3 doses of neoadjuvant cetuximab
  Interventions: Procedure: head and neck surgery

INTERVENTIONS:
Procedure: head and neck surgery — Blood Sample of biomakers at 3 days, 5 weeks and 3 months after surgery.

SUMMARY:
The obvious hypothesis is that the application of peri-operative targeted biological agents may counteract the tumor growth effect of these circulating factors and improve patient outcome

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over

  _ histological proven squamous cell carcinoma of the oral cavity, oropharynx, hypopharinx or larynx
* Patients selected for a primary surgical treatment
* no distant metastases
* no active second malignancy during the last 5 years except non melanoma skin cancer or carcinoma in situ of the cervix
* no prior or concurrent evidence of uncontrolled severe pathology precluding administration of surgery
* life expectancy of more than 3 months
* not pregnant or nursing; fertile patients both male and female, must use effective contraception
* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* signed informed consent
* performance status ECOG 0-1

Exclusion Criteria:

* Nasopharynx cancer
* past or current malignancy other than HNSCC
* performance ECOG status more than 2
* concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
* use of any investigational agents within 4 weeks prior to entry
* Previous exposure to EGFR targeting therapy
* known grade hypersensitivity to cetuximab
* legal incapacity or limited legal capacity or medical or psychological condition which in the opiniion of the investigator would not permit the patient to complete the study or sign meaningful informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
identification of the biomarkers could lead to the development of peri-operative targeted therapies to decrease the risk of local and distant tumor growth | 5 months

SECONDARY OUTCOMES:
Compare the results of group I with groups II and III | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Machiels, PhD, Principal Investigator — Cliniques Universitaires St Luc-UCL
Locations (1):
- Jean-Pascal Machiels, Brussels, Belgium